CLINICAL TRIAL: NCT06776926
Title: When Should Carbetocin be Administered to Prevent Postpartum Hemorrhage After Normal Vaginal Delivery?
Brief Title: Timing of Carbetocin Administration in Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Mete Kırlangıç (Other Government)
Responsible Party: Sponsor-Investigator, Mehmet Mete Kırlangıç, Dr. Lütfi Kırdar Kartal Eğitim ve Araştırma Hastanesi, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Organization: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/514/258/20
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Postpartum Hemorrhage; Carbetocin
Keywords: Postpartum hemorrhage; PPH; Carbetocin; Placental retention
MeSH Terms: conditions — Postpartum Hemorrhage; Placenta, Retained | interventions — carbetocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- After placenta is delivered (Experimental): The group that received carbetocin after placenta delivery
  Interventions: Behavioral: Carbetocin
- Before placenta is delivered (Experimental): The group that received carbetocin before placenta delivery
  Interventions: Behavioral: Carbetocin

INTERVENTIONS:
Behavioral: Carbetocin — Use of carbetocin

SUMMARY:
Postpartum haemorrhage (PPH) is one of the major contributors to maternal mortality and morbidity worldwide. Active management of the third stage of labour has been proven to be effective in the prevention of PPH. Syntometrine is more effective than oxytocin but is associated with more side effects. Carbetocin, a long-acting oxytocin agonist, appears to be a promising agent for the prevention of PPH. The use of carbetocin, being an important agent in the prevention of PPH, also increases its prevalence. It is planned to investigate the advantages and disadvantages of the timing of its use.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Vaginal delivery at or beyond 38 weeks of gestation
* Primipar

Exclusion Criteria:

* Multiparity
* Contraindications to carbetocin use (e.g., pre-existing hypertension, pre-eclampsia,asthma, cardiac, renal, or liver disease)
* High-risk factors for primary postpartum hemorrhage, including grand multiparity,presence of uterine fibroids, or a need for prophylactic oxytocin infusion
* Anemia or
* body mass index (BMI) over 35
* Baby weight over 4000 grams
* Comorbidities or chronic diseases
* History of curettage
* Use of propess or oxytocin during labor

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Carbetosin effect | 24 hours after delivery
  incidence of postpartum hemorrhage >500 ml (percent (%)), additional uterotonics using (yes/no), placenta retention (yes/no), adverse effects (hypotension (yes/no), tachycardia (yes/no), headache(yes/no) oliguria (yes/no)),

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lutfi Kirdar City Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Su LL, Chong YS, Samuel M. Carbetocin for preventing postpartum haemorrhage. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD005457. doi: 10.1002/14651858.CD005457.pub4. PMID 22513931
- [Background] Maged AM, El-Goly NA, Turki D, Bassiouny N, El-Demiry N. A systematic review and meta-analysis of randomized trials comparing carbetocin to oxytocin in prevention of postpartum hemorrhage after cesarean delivery in low-risk women. J Obstet Gynaecol Res. 2025 Jan;51(1):e16194. doi: 10.1111/jog.16194. PMID 39722234
- [Background] Jin B, Du Y, Zhang F, Zhang K, Wang L, Cui L. Carbetocin for the prevention of postpartum hemorrhage: a systematic review and meta-analysis of randomized controlled trials. J Matern Fetal Neonatal Med. 2016;29(3):400-7. doi: 10.3109/14767058.2014.1002394. Epub 2015 Sep 4. PMID 25579116